CLINICAL TRIAL: NCT04460261
Title: The Effects of a New Integrated Exercise Program Called 'Functional' Inspiratory Muscle Training in Geriatric Individuals With and Without Chronic Obstructive Pulmonary Disease
Brief Title: The Effects of 'Functional' Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ismail OZSOY (Other)
Responsible Party: Sponsor-Investigator, Ismail OZSOY, İsmail ÖZSOY, Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20201987
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Exercise
Keywords: chronic obstructive pulmonary disease; functional inspiratory muscle training; geriatric individuals
MeSH Terms: conditions — Motor Activity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and experimental study. The participants were divided into two groups as geriatric individuals with and without chronic obstructive pulmonary disease (COPD). Both groups were trained 3 days a week under the supervision of a physiotherapist and other days of the week without a supervisor. The treatment program consisted of 4 weeks of foundation IMT followed by 4 weeks of functional IMT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD Group (Experimental): Patients with COPD
  Interventions: Other: Functional Inspiratory Muscle Training
- Non-COPD Group (Experimental): Non-COPD
  Interventions: Other: Functional Inspiratory Muscle Training

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training — Both groups were trained 3 days a week under the supervision of a physiotherapist and other days of the week without a supervisor. The treatment program consisted of 4 weeks of foundation IMT followed by 4 weeks of functional IMT. Foundation IMT was applied during the first 4 weeks of training. The participants were asked to sit in a comfortable upright position. Following the foundation IMT, all participants underwent four weeks of functional IMT. Initially, all participants were taught diaphragmatic breathing and activating abdominal wall musculature. Each training session started with warm-up exercises and ended with cool-down exercises. During the loading phase, core stability, dynamic trunk activation and postural control exercises were applied together with IMT.

SUMMARY:
This study was designed as a prospective and experimental study. Geriatric individuals (age ≥ 65 years) with COPD and non-COPD were included in the study. Training program was identical for both groups and consisted of 4 weeks of foundation IMT followed by 4 weeks of functional IMT. Respiratory muscle strength, symptoms, exercise capacity, balance, postural control, physical activity and quality of life were evaluated.

DETAILED DESCRIPTION:
The incidence of chronic obstructive pulmonary disease (COPD), which is one of the most important causes of worldwide mortality and morbidity, increases with age and the disease worsens with the effects of aging. The effects of COPD are not only limited to the lungs, it also affects other organs and systems, causing loss of strength in the respiratory muscles. Respiratory muscles are the skeletal muscles that must maintain their continuous activities for the continuity of life. Just like other skeletal muscles, the respiratory muscles can also be trained based on the principles of exercise. Inspiratory muscle training (IMT) is an exercise method used in both patients with COPD and the elderly population. Studies have shown that IMT has positive effects in COPD and elderly individuals. However, in all these studies IMT applications (also known as "foundation or conventional IMT") focus only on the respiratory task of the respiratory muscles. Nevertheless, in addition to their basic task of respiration, respiratory muscles are also involved in core stabilization and postural control.The aim of this study was to create an integrated IMT program for geriatric individuals with and without COPD and investigate its effects.

The participants were divided into two groups as individuals with and without COPD. A total of 8 weeks of IMT was applied for both groups using a threshold pressure loading device The participants were asked to perform IMT twice a day in the morning and evening. Both groups were trained 3 days a week under the supervision of a physiotherapist and other days of the week without a supervisor. The treatment program consisted of 4 weeks of foundation IMT followed by 4 weeks of functional IMT.The intensity of the exercise was adjusted to 40-50% of the MIP. After 10 consecutive breathing cycles, the participants were asked to perform 3-4 breathe controls. As the tolerance increased, consecutive respiratory cycles were increased. The intensity of MIP was adjusted by weekly MIP measurements. Currently, foundation IMT is commonly used to train respiratory muscles. In the present study, foundation IMT was applied during the first 4 weeks of training. The participants were asked to sit in a comfortable upright position. Then the nose clip was placed, and the patients were instructed to tighten their lips around the mouthpiece and breathe against the resistance. During this 4-week-long training, all IMT applications were performed solely in a sitting position, without any loading in other positions. Following the foundation IMT, all participants underwent four weeks of functional IMT. Initially, all participants were taught diaphragmatic breathing and activating abdominal wall musculature. Each training session started with warm-up exercises and ended with cool-down exercises. During the loading phase, core stability, dynamic trunk activation and postural control exercises were applied together with IMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing COPD in accordance with Global initiative for chronic obstructive pulmonary disease (GOLD) guideline criteria
* Being over 65 years old
* Being a stable clinical condition (same medication routine for the past 3 weeks without taking any antibiotics)
* Independent mobilization
* Note: Normal spirometry values set as the inclusion criteria for non-COPD group.

Exclusion Criteria:

* Orthopaedic problems
* Neurological problems
* Cognitive problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 8 weeks
  Inspiratory muscle strength (MIP) was measured using a hand-held mouth pressure device (Micro RMP; Micro Medical, Rochester, UK). Three to five acceptable and reproducible maximal manoeuvres (i.e., differences between values <10%) were performed and the highest value was recorded.
Expiratory muscle strength | 8 weeks
  Expiratory muscle strength (MEP) was measured using a hand-held mouth pressure device (Micro RMP; Micro Medical, Rochester, UK). Three to five acceptable and reproducible maximal manoeuvres (i.e., differences between values <10%) were performed and the highest value was recorded.
Dyspnea assessment | 8 weeks
  The Modified Medical Research Council (mMRC) Dyspnea Scale was used to evaluate dyspnea. Commonly used in the assessment of dyspnea in COPD, mMRC has a five-level scoring system ranging from 0 to 4. A high score indicates an increased sense of dyspnea.
Symptoms assessment | 8 weeks
  The COPD Assessment Test (CAT) was used to assess symptoms in patients with COPD. It is a reliable test to evaluate the impact of COPD on a patient's health status. It has eight items and the score ranges from 0 to 40. Higher scores indicate increased symptoms.
Upper extremity functional exercise capacity assessment | 8 weeks
  The 6-Minute Pegboard and Ring Test was used to assess upper extremity functional exercise capacity assessment
Lower extremity functional exercise capacity assessment | 8 weeks
  The 6-Minute Walking Test (6MWT) was used to assess lower extremity functional exercise capacity assessment.

SECONDARY OUTCOMES:
Balance assessment | 8 weeks
  Balance was assessed using Berg Balance Scale (BBS). This scale consists of 14 items and each item is scored between 0 and 4. A higher score indicates better balance.
Static antero-posterior postural stability assessment | 8 weeks
  A portable balance device (Biodex Biosway Portable Balance System, New York, USA) was used to measure static antero-posterior postural stability.A higher score indicates a lower level of postural control.
Static medio-lateral postural stability assessment | 8 weeks
  A portable balance device (Biodex Biosway Portable Balance System, New York, USA) was used to measure static medio-lateral postural stability. A higher score indicates a lower level of postural control.
Physical activity assessment | 8 weeks
  Physical activity was assessed using the Physical Activity Scale for the Elderly (PASE). It is a validated 12-item self-administered scale in which higher scores indicate increased physical activity.The overall PASE score ranges from 0 to 400 or more and high scores show better physical activity levels.
Quality of life assessment | 8 weeks
  The quality of life was assessed using the World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD). This questionnaire consists of 24 items in six different domains and higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail ozsoy, PhD, Principal Investigator — Selcuk University